CLINICAL TRIAL: NCT06882538
Title: The Effect of Mindfulness-Based Psychoeducation Programme Given Individually to Schizophrenia Patients on Internalised Stigma and Healthy Lifestyle Behaviours
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kastamonu University (Other)
Responsible Party: Principal Investigator, Havva Kaçan, ASSOCIATE PROFESSOR, Kastamonu University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024/20/4; 2024/20/4 (Other: Kastamonu University)
Record Dates: First submitted 2025-02-14; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-02

CONDITIONS: Schizophrenia Disorders
Keywords: schizophrenia; psychoeducation; internalised stigmatisation; healthy lifestyle behaviour
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: Patients who were followed up at Kastamonu University Training and Research Hospital Community Mental Health Centre between April 2024 and May 2024 with a diagnosis of schizophrenia according to DSM-5 diagnostic criteria will be included in the study. All patients will be informed about the nature of the interview and scales and written informed consent will be obtained from patients who accept the evaluation. Written permission will be obtained from the Provincial Directorate of Health for the study. The study group patients will be divided into two groups and the training will be given in 12 sessions as two lessons of forty-five minutes each once a week and will be completed in approximately 6 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Awareness-Based Psychoeducation (Experimental): Sessions
  1. Meeting with the group members, introduction of the group process, explanation of the session topics,
  2. Information about the management of schizophrenia
  3. Information about the management of schizophrenia
  4. Taking Responsibility in Health,
  5. Gaining Positive Health Behaviours: Nutrition and Exercise, Hygiene practices skills training
  6. Gaining Positive Health Behaviours: Using Interpersonal Communication and Supports, Anger Management
  7. Acquiring Positive Health Behaviours: Self-actualisation,
  8. Gaining Positive Health Behaviours: Managing Stress,
  9. Gaining Positive Health Behaviours: Managing Stress, Progressive relaxation techniques
  10. Dealing with stigmatisation
  11. Dealing with stigmatisation
  Interventions: Other: awareness-based psychoeducation

INTERVENTIONS:
Other: awareness-based psychoeducation — The aim of psychoeducation is to create a change in knowledge and behaviour towards healthy lifestyle behaviours (1- Self-actualisation, 2- Health responsibility, 3- Exercise, 4- Nutrition, 5- Interpersonal support, 6- Stress management) by reducing internalised stigma. Therefore, it will be evaluated whether the applied psychoeducation programme creates the intended change in knowledge and behaviour.

SUMMARY:
Schizophrenia is a chronic, recurrent and disabling illness that usually lasts a lifetime and causes serious problems in quality of life and functioning. Psychoeducation programmes added to drug treatment in the treatment of schizophrenia have been shown to increase the knowledge of patients and their relatives about the disease, coping skills, prevention of exacerbations and relapses of the disease, social functioning, insight into the disease, compliance with drug treatment and quality of life. Rehabilitated individuals diagnosed with schizophrenia who are registered and continuing at Kastamonu Training and Research Community Mental Health Centre will constitute the population, and individuals who continue between April 2024 and May 2024 will constitute the sample. The research will be conducted with schizophrenic patients in a pre-test-post-test, experimental and control group experimental design. Power analysis will be performed to determine the number of people to be sampled and calculated with the G*Power 3.1 programme. 40 people will be reached in the groups, 20 people in the experimental group and 20 people in the control group. In the evaluation of the data, descriptive statistical methods (Mean, Standard deviation) as well as the correlation test will be used to evaluate the relationship between the average scores before and after the training in the comparison of quantitative data. Wilcoxon related sample test will be used to make comparisons before and after the training. Personal Information Form, Internalised Stigma Scale in Mental Illness (ISIS) and Healthy Lifestyle Behaviours (HBSB) scale will be used to collect the data. Awareness-based psychoeducation programme will be applied to the experimental group. The aim of psychoeducation is to create a change in knowledge and behaviour towards healthy lifestyle behaviours (1- Self-actualisation, 2- Health responsibility, 3- Exercise, 4- Nutrition, 5- Interpersonal support, 6- Stress management) by reducing internalised stigma. Therefore, it will be evaluated whether the applied psychoeducation programme creates the intended change in knowledge and behaviour. This study will be conducted to examine the effect of a 6-week 12-session self-awareness-based psychoeducation programme given to schizophrenia patients on internalised stigma and healthy lifestyle behaviours. In this study, schizophrenic patients will be provided with regular psychoeducation to provide individual support, to ensure the development of coping skills for self-protection, and to gain knowledge and skills to gain a healthy lifestyle. After the prepared psychoeducation, a training guide will be created for the participants and will be given after the training, thus ensuring continuity of education.

DETAILED DESCRIPTION:
Research Population/Sample or Study Group: If appropriate in terms of the study method, the population and sample should be explained here. Specify how the sample/study group will be selected, how they will be assigned to groups and which sampling method(s) (e.g. random-probability, snowball, convenience, purposive, cluster sampling) will be used.

Rehabilitated individuals diagnosed with schizophrenia who are registered and attending the Community Mental Health Centre will constitute the population, and individuals attending between April 2024 and May 2024 will constitute the sample. Power analysis will be performed to determine the number of people to be sampled and calculated with the G*Power 3.1 programme. In the literature, while there is an interventional study on stigmatisation among similar interventional studies for previously diagnosed schizophrenic patients, there is no study investigating stigmatisation and healthy lifestyle behaviours. The effect size was taken as 0.80 as a high level according to the t-test determined by Cohen (1988). In order to exceed the 95% value in determining the power of the study; 40 people, including 20 people in groups with a significance level of 5% and an effect size of 0.80, should be reached (df=68; t=1.668). Since the training covers a period of 6 weeks, schizophrenic individuals who are willing and will continue the training will be accepted.

Data Collection Tool:

Personal Information Form, Internalised Stigma Scale in Mental Illness (ISIS) and Healthy Lifestyle Behaviours (HBSB) scale will be used to collect the data.

Internalised Stigma Scale in Mental Illness (ISIS): Developed by Ritsher et al. (2003), RHIAS is a self-report scale consisting of 29 items and assessing internalised stigma . Turkish adaptation study was conducted by Ersoy and Varan 6. RHIDÖ is a four-point Likert-type scale. The scale has five subscales; 1. Alienation, 2. Confirmation of Stereotypes, 3. Perceived Discrimination, 4. Social Withdrawal and 5. Resistance to Stigmatisation. The items of the 'Resistance to Stigmatisation' subscale are reverse scored.

Total score varies between 29 and 116 points. High scores obtained from the RHIDÖ indicate a high level of internalised stigma. In Ersoy and Varan's study, the Cronbach Alpha value of the scale was 0.93. The scale has been authorised for use and is available in the appendices.

Healthy Lifestyle Behaviours (HLSB) Scale: Developed in 1987 by Walker, Sechrist and Pender, the HLSBS measures the health-promoting behaviours of the individual in relation to healthy lifestyle. It was adapted into Turkish by Esin, a validity and reliability study was conducted and Cronbach's Alpha internal consistency coefficient was found to be 0.91. The scale is a four-point Likert-type scale consisting of a total of 48 items and six subgroups. The score of each subgroup of the scale can be used alone or the total score of the whole scale can be used and gives the score of healthy lifestyle behaviours. The highest score for the whole scale is 192 and the lowest score is 48. A high score on the scale indicates better healthy lifestyle behaviours. All items of the scale are positive and there is no reverse-scored item. The subgroups of the scale are as follows: Self-actualisation; It consists of a total of 13 items covering 3, 8, 11, 12, 16, 17, 21, 23, 29, 34, 37, 44 and 48 questions. It determines the individual's life goals, individual self-development ability, and the extent to which he/she recognises and satisfies himself/herself. Health responsibility consists of a total of 10 items (2, 7, 15, 20, 20, 28, 32, 33, 42, 43 and 46). It determines the level of responsibility of the individual on his/her own health and the extent to which he/she participates in his/her health. Exercise; shows the level of exercise, which is an unchangeable element of healthy life, and consists of a total of 5 items (4, 13, 22, 30 and 38). Nutrition; It consists of a total of 6 items covering 1, 5, 14, 19, 26 and 35 questions. It determines the individual's values in choosing and organising meals and choosing food. Interpersonal support determines the communication and continuity level of the individual with his/her close environment and consists of 7 items (10, 18, 24, 25, 31, 39, and 47). Stress management consists of a total of 7 items (6, 9, 27, 36, 40, 41, and 45) that determine the individual's level of recognition of stress sources and stress control mechanisms.

Data Collection Process: The data will be collected by face-to-face interview method by the researchers. It will be done within the knowledge of the institutional staff within the time interval when they come to the community mental health centre. Pre-test applications will be made to individuals before psychoeducation is given. 6-week training will be given to individuals one by one. Each individual will be provided with 6 weeks of training. After the training, data collection tools will be applied again and post-tests will be created. 20 individuals will be included in the experimental group and 20 individuals will be included in the control group.

ELIGIBILITY:
Inclusion Criteria:

1. Having been diagnosed with schizophrenia
2. TRSM registered and continuing
3. Acceptance to work and training

Exclusion Criteria:

1. Have not been diagnosed with schizophrenia
2. If he/she does not agree to participate in the study
3. If not registered with TRSM

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
The level of internalized stigma of schizophrenia patients | Four Week
  In this study, the level of internalized stigma in schizophrenia patients will be measured with the internalized stigma scale.

SECONDARY OUTCOMES:
Healthy lifestyle behaviors of schizophrenia patients participating in psychoeducation will be evaluated. | Four Week
  The frequency of healthy lifestyle behaviors of schizophrenia patients receiving psychoeducation will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Havva K KAÇAN, ASSOCIATE PROFESSOR DOCTOR, Principal Investigator — Kastamonu University
Locations (1):
- Kastamonu Community Mental Health Centre, Kastamonu, Central, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided